CLINICAL TRIAL: NCT04091802
Title: Effect of Monolayer Versus Multilayer Leucocyte-Platelet Rich Fibrin (L-PRF) in Interdental Papillary Reconstruction" (A Randomized Controlled Clinical Study)
Brief Title: Effect of Monolayer Versus Multilayer Leucocyte-Platelet Rich Fibrin (L-PRF) in Interdental Papillary Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Amir ahmed Lashin, Principle investigator at Ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECO 1214403
Record Dates: First submitted 2019-08-27; First posted 2019-09-17 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Recession
Keywords: interdental papilla reconstruction; Leucocyte-Platelet Rich Fibrin (L-PRF)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single layer of L-PRF (Experimental): single layer of L-PRF will be put in the vertical incision
  Interventions: Procedure: interdental papilla reconstruction with L-PRF
- multiple layers of L-PRF (Experimental): multiple layers of L-PRF will be put in the vertical incision
  Interventions: Procedure: interdental papilla reconstruction with L-PRF

INTERVENTIONS:
Procedure: interdental papilla reconstruction with L-PRF — interdental papilla reconstruction with single layer of L-PRF versus multiple layers of L-PRF

SUMMARY:
The interdental papilla is very small but it has a great implication from an aesthetic view, more specifically in the anterior region because it is always displayed during smiling. The lack of interdental papilla due to periodontal disease or periodontal therapy leads to aesthetic problems with food stagnation as well as phonetic problem due to the space that allows passage of the air or saliva. Leukocyte-PRF (L-PRF) membrane was developed which includes the majority of the platelets in addition to half of the leukocytes so that lymphocytes as well as the platelet growth factors are trapped inside a fibrin network. Multiple layers of L-PRF may have observable effect on tissue regeneration because it increases the number of growth factors and acts as a strong scaffold which helps in creeping of the cells along it as it remains active and in place for more than 7 days. Thus, the aim of this study will be conducted to compare the effect of one layer versus multiple layers of L-PRF in interdental papillary reconstruction.

DETAILED DESCRIPTION:
A total of 20 patients will be selected who are caring about esthetics and concerned to go through the management of eradication of "black triangles" by interdental papillae reconstruction in esthetic zone and systemically free with Nordland's class I or II and The vertical distance from the interdental contact point to the crest of the interdental bone is ≥ 6 mm as measured by bone sounding, A band of keratinized tissue should be present around the test teeth ≥ 2 mm, Gingival biotype of the area to be treated is ≥ 2 mm in thickness.

The study protocol will be explained in details to all patients. Then a signed informed consent will be obtained from the patients. The data obtained from patients as well as the results of the follow up will be kept confidential.

The study will be introduced to ethics' committee of Faculty of Dentistry Ain Shams University and has to be approved before the start of the study Eligible patients will be randomized in a 1:1 ratio into two groups; (Group I) included 10 patients and (Group II) included 10 patients. The computer-generated randomization assignment (blocks of 4) and allocation concealment will be performed by sealed envelopes containing the randomization number prepared by non involved member and sent to principle investigator to assign the interventions to patients Group I: 10 patients will undergo interdental papillary reconstruction using one layer of L-PRF.

Group II: 10 patients will receive interdental papillary reconstruction using multiple layers of L-PRF (Two or more according to the compressibility in which if ≥1mm, it needs one more layer, and if ≤1 mm, then no need to more than 2 layers; it cannot be standardized).

Procedure:

1. All patients will receive Phase I therapy including oral hygiene measures and scaling and root planning whenever indicated.
2. Preparation of recipient site:

   The preparation of the recipient site is similar to that described by Reddy.
   * Anasthesia of the surgical field.
   * A single vertical incision will be made in the buccal vestibule apical to the mucogingival junction in the mid interproximal area of the papilla to be treated.
   * Intrasulcular releasing incisions will be made on the teeth adjacent to the papilla to be augmented and extend to the buccal and palatal aspects without altering the integrity of the papilla.
   * The incisions will maintain the full height and thickness of the gingiva.
   * Papilla will be undermined carefully to maintain integrity and a space will be created under the papilla by elevating it coronally.
3. Preparation of L-PRF:

   L-PRF will be prepared according to Chaukroun's et al. 2001. Immediately prior to the surgery, 10 ml of blood (for each membrane) will be collected from the patient by venipuncture of antecubital vein and then drawn quickly into sterile glass tube with no anticoagulant and immediately centrifuged at 2700 rpm for 12 minutes at room temperature by using the Intra-Spin centrifuge (Intra-Lock).

   Then L-PRF clot will be removed by sterile tweezers and placed in Xpression™ kit for gentle compression by gravity. Then L-PRF will be ready to be used after 5 minutes (For group II, membranes will be sutured together before placement in the vertical incision).
4. Placement and suturing of L-PRF in the recipient site:

   The L-PRF membrane will be trimmed to the desired shape and size and then placed under the papilla and mucogingival complex through the vertical incision to fill the black space.

   Then incision will be closed with 5-0 polypropylene simple interrupted sutures.
5. Post operative management:

It will include pain control using anti-inflammatory and analgesics (Brufen 600 mg) when needed and twice mouth rinse with chlorohexidine gluconate daily for one week.

All Clinical and volumetric measurements will be carried out at baseline and after 6 months follow up and esthetic assessment will be done.

Clinical assessment will be Plaque score index (PI), gingival score index (GI), papillary height from the tip of the papilla to mesial line angle, Nordland and Tarnaw classification.

volumetric assessment will be with intraoral scan with CAD-CAM preoperative and 6 months postoperative.

Esthetic assessment will be done by means of the root coverage esthetic score (RES), this score estimates five variables: gingival margin level (GM), the contour of the marginal tissue (MTC), soft tissue texture (STT), location of mucogingival junction (MGJ), and gingival color (GC). Zero, 3, or 6 points will be used for the estimation of the location of the gingival margin, while a score of 0 or 1 point will be used for each of the other variables.GM. Zero points = no root coverage (in which the gingival margin is in equal level to the baseline or migrated apically); 3 points = partial coverage; 6 points = Complete coverage.

MTC. Zero points = asymmetrical gingival margin (does not track the CEJ); 1point = appropriate marginal contour/ scalloped gingival margin (tracks the CEJ).

STT. Zero points = scar development; 1 point = absence of scar. MGJ. Zero points =MGJ is not uniform with the MGJ of neighboring teeth; 1 point = MGJ is uniform with the MGJ of neighboring teeth.

GC. Zero points = tissue color differs from gingival color of neighboring teeth; 1 point = normal color and unification with the neighboring soft tissues.

Accordingly, the perfect esthetic score is 10. Satisfaction questionnaire, to score degree of pain experienced during and after treatment and the degree of patient satisfaction with the cosmetic results of the procedure.

All data will be collected blindly and subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed with black triangles. 2. Both genders aged from 18-40 years. 3. Patients should be systemically free. 4. Patients with Nordland's class I or II. Nordland and Tarnow classified the interdental papilla loss; the classification is based on three anatomic landmarks: the contact point interdentally, the coronal level of the CEJ interproximally and the facial apical level of the cemento-enamel junction (CEJ). [Nordland WP, et al, 1998] Four classes were identified

  * Normal: The interdental papilla fills up the whole embrasure to the interproximal contact point.
  * Class I: Presence of the tip of the papilla between interdental contact point and the interproximal CEJ.
  * Class II: Presence of the tip of the papilla at the interproximal CEJ or apical to it but still coronal to the facial CEJ.
  * Class III: Presence of the tip of papilla at similar plane with the labial CEJ or apical to it.

    5. The vertical distance from the interdental contact point to the crest of the interdental bone is ≥ 6 mm as measured by bone sounding.

    6. A band of keratinized tissue should be present around the test teeth ≥ 2 mm. 7. Gingival biotype of the area to be treated is ≥ 2 mm in thickness.

Exclusion Criteria:

1. Acute periapical lesion.
2. moderate to severe form of periodontitis.
3. Pregnancy and lactation.
4. parafunctional habits.
5. Smoking, alcoholics or drug abusers.
6. Teeth with interdental spacing, rotation or inclination or crowding.
7. Vulnerable group of patients.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
clinical assessment | change from baseline to 6 months
  papillary height from the tip of the papilla to mesial line angle

SECONDARY OUTCOMES:
volumetric analysis | change from baseline to 6 months
  intraoral scan with CAD-CAM

CONTACTS AND LOCATIONS:
Overall Officials: Nivine H. kheir el den, professor, Study Chair — faculty of dentistry- ain shams university

IPD SHARING:
Plan to Share IPD: No